CLINICAL TRIAL: NCT01375907
Title: A Phase 1 Study to Evaluate Safety and Reactogenicity of a Vietnamese Rotavirus Vaccine (Rotavin-M1 at 10e6.3FFU/Dose) Among Healthy Adults in Vietnam
Brief Title: Safety Study of a Rotavirus Vaccine (Rotavin-M1) Among Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Center for Research and Production of Vaccines and Biologicals (Unknown)
Responsible Party: Principal Investigator, Dang Duc Anh, Director, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Rotavin01
Record Dates: First submitted 2011-05-19; First posted 2011-06-17 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Diarrhea; Vomit; Fever; Nausea; Irritability
Keywords: blood cell counts; BUN; ALT; AST; diarrhea; fever; vomit; nausea; loss of appetite; irritability
MeSH Terms: conditions — Diarrhea; Vomiting; Fever; Nausea; Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rotavin (Experimental): Rotavin-M1 vaccine, 10e6.3FFU/dose, 2 doses, 1 month between doses
  Interventions: Drug: Rotavin

INTERVENTIONS:
Drug: Rotavin — Rotavin-M1, 10e6.3FFU/dose, 2 doses, 1-month between doses
  Other Names: Rotavin-M1

SUMMARY:
The purpose of this study is to evaluate the safety of Rotavin-M1 produced by the Center for Research and Production of Vaccines and Biologicals (POLYVAC) in adult volunteers in Vietnam.

DETAILED DESCRIPTION:
Rotavirus (RV) is the most important cause of acute gastroenteritis in children worldwide. In Vietnam rotavirus causes an estimated 122,000-140,000 hospitalizations and 2900-5400 deaths per year among children under 5 years of age (1). Over the past 13 years, sentinel hospital surveillance identified rotavirus in 44%-62% of children admitted for the treatment of acute diarrhea in Vietnam (2-4). Such a high burden of disease justified accelerated development of a new and locally manufactured vaccine against rotavirus in Vietnam. It is estimated that if a vaccine was introduced in the current childhood immunization schedule, it could reduce severe rotavirus disease by about 60% or more given current vaccine efficacies and coverage (5).

The Government of Vietnam has pursued a policy to encourage local vaccine production so the country could be self-reliant with affordable vaccines for its population (6). Over the past decades, several locally produced vaccines for poliomyelitis, cholera, Japanese encephalitis, and Diphtheria-Pertussis-Tetanus have contributed to the reduction in the prevalence of these diseases and to the eradication of polio over the past decade. While two commercial rotavirus vaccines, RotarixTM (GSK, Belgium) and RotaTeq® (Merck), have both been tested in Vietnam, neither is currently available at an affordable cost for the national program. Therefore, the candidate vaccine, Rotavin-M1, was developed in order to fill this need for a more affordable vaccine for Vietnamese children (6). This vaccine is similar to RotarixTM, and was developed by selecting a common G1P[8] strain and attenuating it through serial

ELIGIBILITY:
Inclusion Criteria:

At dose 1

* Healthy male or female, 18 to 40 years of age,
* Free of disease,
* Written informed consent obtained from subjects. At dose 2
* Received dose 1.
* Oral informed consent obtained from subject for continuing participate the study.

Exclusion Criteria:

At dose 1

1. Pregnant woman or planning to be pregnant during the study period.
2. Has a chronic disease (cardiovascular, liver, kidney disease).
3. Acute disease at the time of enrolment.
4. Administering corticosteroids (> 1mg/kg/day).
5. Received any immunosuppressive therapy within 4 week before vaccination (Administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
6. Immunosuppressive or immunodeficient condition.
7. Allergic or reaction with any component of vaccine, includes anaphylactic and shock with any antibiotic.
8. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
9. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
10. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine during the study period.

At dose 2

1. Pregnant woman or planning to be pregnant in next 1 month.
2. Acute disease at the time of 2nd dose.
3. Administering corticosteroids (> 1mg/kg/day).
4. Received any immunosuppressive therapy within 4 week before vaccination (administration of immunoglobulins and/or any blood product or corticosteroids for >2 weeks).
5. Immunosuppressive or immunodeficient condition.
6. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
7. Fever (axillary temperature >38oC) within 3 days before or on the day of vaccination.
8. Has any type of blood disorder, leukemia, or malignant tumor which can affect the bone marrow or lymph system.
9. Use of any investigational or non-registered product (unlicensed drug or vaccine) other than the study vaccine during the study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety of Rotavin-M1 vaccine in healthy adult volunteers | 3 months
  To evaluate the safety of 2 doses Rotavin-M1 vaccine (10e6.3FFU/dose, 1-month interval between doses) in healthy adult volunteers.

SECONDARY OUTCOMES:
Reactogenicity of Rotavin-M1 in healthy adult volunteer | 3 months
  To evaluate immediate reactions (30 minutes) after administration of each dose
Change in blood cell counts, serum transaminase and urea nitrogen concentration in adults after vaccination with Rotavin-M1 | 3 months
  to assess change in blood cell counts (red blood cells, white blood cells, platelets), blood urea nitrogen concentration, serum transaminase levels (AST, ALT) in adult volunteer after each dose of Rotavin-M1 10e6.3FFU/dose

CONTACTS AND LOCATIONS:
Overall Officials: Anh D Dang, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (1):
- Preventive Medicine Center, Thanh Sơn, Phu Tho, Vietnam

REFERENCES:
- [Background] Anh DD, Thiem VD, Fischer TK, Canh DG, Minh TT, Tho le H, Van Man N, Luan le T, Kilgore P, von Seidlein L, Glass RI. The burden of rotavirus diarrhea in Khanh Hoa Province, Vietnam: baseline assessment for a rotavirus vaccine trial. Pediatr Infect Dis J. 2006 Jan;25(1):37-40. doi: 10.1097/01.inf.0000195635.05186.52. PMID 16395100
- [Background] Van Man N, Luan le T, Trach DD, Thanh NT, Van Tu P, Long NT, Anh DD, Fischer TK, Ivanoff B, Gentsch JR, Glass RI; Vietnam Rotavirus Surveillance Network. Epidemiological profile and burden of rotavirus diarrhea in Vietnam: 5 years of sentinel hospital surveillance, 1998-2003. J Infect Dis. 2005 Sep 1;192 Suppl 1:S127-32. doi: 10.1086/431501. PMID 16088796
- [Background] Ngo TC, Nguyen BM, Dang DA, Nguyen HT, Nguyen TT, Tran VN, Vu TT, Ogino M, Alam MM, Nakagomi T, Nakagomi O, Yamashiro T. Molecular epidemiology of rotavirus diarrhoea among children in Haiphong, Vietnam: the emergence of G3 rotavirus. Vaccine. 2009 Nov 20;27 Suppl 5:F75-80. doi: 10.1016/j.vaccine.2009.08.074. PMID 19931725
- [Background] Nguyen TA, Yagyu F, Okame M, Phan TG, Trinh QD, Yan H, Hoang KT, Cao AT, Le Hoang P, Okitsu S, Ushijima H. Diversity of viruses associated with acute gastroenteritis in children hospitalized with diarrhea in Ho Chi Minh City, Vietnam. J Med Virol. 2007 May;79(5):582-90. doi: 10.1002/jmv.20857. PMID 17385670
- [Background] Kim SY, Goldie SJ, Salomon JA. Cost-effectiveness of Rotavirus vaccination in Vietnam. BMC Public Health. 2009 Jan 21;9:29. doi: 10.1186/1471-2458-9-29. PMID 19159483
- [Background] Luan le T, Trang NV, Phuong NM, Nguyen HT, Ngo HT, Nguyen HT, Tran HB, Dang HN, Dang AD, Gentsch JR, Wang Y, Esona MD, Glass RI, Steele AD, Kilgore PE, Nguyen MV, Jiang B, Nguyen HD. Development and characterization of candidate rotavirus vaccine strains derived from children with diarrhoea in Vietnam. Vaccine. 2009 Nov 20;27 Suppl 5:F130-8. doi: 10.1016/j.vaccine.2009.08.086. PMID 19931712
- [Derived] Dang DA, Nguyen VT, Vu DT, Nguyen TH, Nguyen DM, Yuhuan W, Baoming J, Nguyen DH, Le TL; Rotavin-M1 Vaccine Trial Group. A dose-escalation safety and immunogenicity study of a new live attenuated human rotavirus vaccine (Rotavin-M1) in Vietnamese children. Vaccine. 2012 Apr 27;30 Suppl 1:A114-21. doi: 10.1016/j.vaccine.2011.07.118. PMID 22520120